CLINICAL TRIAL: NCT00675389
Title: Impact of Peer Health Workers and Mobile Phones on HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Doris Duke Charitable Foundation (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Larry William Chang, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00000748
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Community Health Workers; Mobile Phones; Adherence; Antiretroviral Therapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Peer Health Workers Intervention
  Interventions: Behavioral: Peer Health Workers Intervention
- B (Experimental): Peer Health Workers and Mobile Phone Intervention
  Interventions: Behavioral: Peer Health Workers and Mobile Phone Intervention
- C (No Intervention): Control

INTERVENTIONS:
Behavioral: Peer Health Workers Intervention — Peer health workers are themselves PLWHA on ART who have demonstrated good ART adherence for at least 6 months. The peers are responsible for ~15-20 patients and are expected to visit the patients in their homes once every two weeks. At these visits, peers record a review of symptoms, client self-report of adherence, and a pill count. At the clinic, peers assist with patient organization and share their experiences, particularly with patients about to start ART. Peer health workers undergo an initial, intensive two day residential training course and are provided with a bike and basic supplies, and a modest amount of remuneration to encourage compliance with their responsibilities and promote a high program retention rate.
  Arms: A
Behavioral: Peer Health Workers and Mobile Phone Intervention — In addition to the peer health worker intervention, this arm adds a mobile phone intervention consisting of the following: during home visits, peers with mobile phones, using data collected on their home visit forms, send real-time text messages containing this clinical and adherence data back to the central clinic to be reviewed by clinical staff within a 24 hour period. Peers may also call, toll-free, back to a central clinic Warmline with any questions or concerns.
  Arms: B

SUMMARY:
The provision of antiretroviral therapy (ART) in rural, resource-limited settings entails substantial challenges due to limitations in the health service infrastructure and in human resources for HIV/AIDS care. In addition, long geographical distances between providers, care facilities, and patients can represent a significant barrier to appropriate and timely care. The use of peer health workers as frontline adherence supporters and clinical monitors in order to improve care in underserviced settings has been implemented by a number of programs, but the effect of peer support on HIV care outcomes has not been extensively evaluated. Mobile phones have also been proposed as a potential method of improving access to health care in resource-limited environments by expediting communication and data transfer, but rigorous studies on their effectiveness in Africa have not yet been conducted.

The Rakai Health Science Project (RHSP) was founded in 1987 to study the HIV epidemic in the rural setting of Rakai District in southwest Uganda. Since June 2004, the US President's Plan for AIDS Relief (PEPFAR) has enabled the RHSP to provide ART through a community-based distribution system which includes clinical monitoring via a decentralized, mobile clinic approach. By late 2006, the program has screened 4,397 HIV-infected individuals and initiated ART in 849 patients. One of the challenges of providing ART in this setting has been the distance between many patients' homes and the clinic and medical staff trained in HIV care. This distance and the lack of communication channels make frequent clinic contacts difficult and has raised concerns about adherence and management of drug toxicity. This study will investigate whether peer health workers can help support this AIDS care program and improve patient outcomes.

This study is a three armed, community-randomized operations research trial to assess the effectiveness of peer health workers, with and without mobile phones, in improving the delivery of HIV care in the resource-limited Rakai setting. The three arms will be: a) communities with peer health workers, b) communities with peer health workers and mobile phones, and c) control communities without peer health workers.

Study hypotheses include:

* Peer health workers, by supporting adherence and by managing simple clinical issues, will reduce virologic treatment failure and improve ARV adherence compared to patients in communities without peer educators.
* Mobile phone technology used by peer health workers, by more rapidly addressing adherence and clinical problems, will reduce treatment failure and improve adherence compared to patients in communities with peer health workers without mobile phones.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the study is determined by receipt of ARVs in the PEPFAR program.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Virologic suppression at 6 months | 6 months
Virologic failure at all time intervals from ART initiation (these primary outcomes added to expanded trial protocol November 2007) | Typically every 24 weeks
Adherence measured by pill counts (this primary outcome added to expanded trial protocol November 2007) | Typically weekly to monthly

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Gray, MBBS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Larry W Chang, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine

REFERENCES:
- [Derived] Chang LW, Kagaayi J, Nakigozi G, Ssempijja V, Packer AH, Serwadda D, Quinn TC, Gray RH, Bollinger RC, Reynolds SJ. Effect of peer health workers on AIDS care in Rakai, Uganda: a cluster-randomized trial. PLoS One. 2010 Jun 2;5(6):e10923. doi: 10.1371/journal.pone.0010923. PMID 20532194